CLINICAL TRIAL: NCT06311162
Title: Early Life Intervention in Pediatrics Supported by E-health (ELIPSE II): Coaching Parents to Lower Second-hand Smoke Exposure in Children A Single-blind Randomized Controlled Parallel-group Clinical Trial
Brief Title: Early Life Intervention in Pediatrics Supported by E-health - SMOKE
Acronym: ELIPSE-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-01615
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Smoking Reduction; Asthma in Children; Wheezing; Non-Communicable Disease; Life Style; Behavior, Smoking
Keywords: Secondhand smoke; Children; Prevention; eHealth
MeSH Terms: conditions — Smoking Reduction; Respiratory Sounds; Noncommunicable Diseases; Smoking

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled parallel-group clinical trial
Who Masked: Care Provider, Investigator
Masking Description: The study team members who are conducting assessments on the participants remain blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Life-style app) (Experimental): Parents receive a smartphone app during the main intervention period of 20 weeks. The app (life-style app) aims to promote healthy behaviour through cognitive-behavioural impact factors.
  Interventions: Behavioral: Life-Style app
- Control group (Sham Comparator): The parents get an information sheet with information on second-hand smoke exposure and references to smoking cessation programs, and do not have an active app during the main intervention period.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Behavioral: Life-Style app — The modules of the Life-Style app are introduced and unlocked sequentially during the first weeks of the intervention phase. Afterwards the modules are fully available. Duration and frequency of app-use is not limited. The parents are accompanied by a coach through the app, who gives regular structured feedback and individual inputs. The coach has access to all data collected in the app.
  Other Names: Smartphone App
  Arms: Treatment group (Life-style app)
Other: Sham Comparator — The parents get a flyer with information on second-hand smoke exposure and references to smoking cessation programs, and do not have an active app during the main intervention period.
  Other Names: Flyer about second-hand smoke exposure
  Arms: Control group

SUMMARY:
Unrestricted parental smoking habits are lifestyle risk behaviors associated with chronic, systemic inflammation, which promotes the pathogenesis of non-communicable diseases (NCDs). Exposure to secondhand tobacco smoke in early life contributes to the development of specific NCDs in children, i.e. asthma. Early preventive measures to improve lifestyle behavior in parents are therefore of utmost importance. The aim of ELIPSE-II is to assess whether an eHealth application intervention for parents is feasible and efficacious in lowering levels of urinary cotinine as a measure of second-hand smoke exposure in their children .

DETAILED DESCRIPTION:
ELIPSE-II represents a single-blind randomized controlled parallel-group clinical trial. In total, 160 children, <6 years of age with exposure to second-hand smoke at home will be included. Children will be recruited at the children's university hospital and in private practices in Bern, and randomly (1:1) assigned to a control and intervention group.

All participants receive treatment-as-usual (TAU), parents of participants in the intervention group additionally receive a smartphone application (lifestyle app) for 20 weeks. The app aims to promote healthy behavior through cognitive-behavioral impact factors (i.e., psychoeducation, goal setting), that are applied by a psychologist via structured feedback. Single-blinded assessments will be conducted at baseline, following the intervention period of 20 weeks, and at 6-month follow-up after the end of the intervention. The primary endpoint is reduction of exposure to second-hand smoke exposure assessed by urinary levels of cotinine. Secondary endpoints in ELIPSE-II include changes in parental smoking habits and effects of the intervention on infants' respiratory health. A further endpoint is acceptance and usability of the app.

ELIGIBILITY:
Inclusion Criteria:

* Age: younger than 6 years
* Exposed to second-hand smoke at home (at least one parent smoking)
* German speaking parent
* All sex and ethnic backgrounds
* Signed informed consent form from parent
* Children live/grow-up in the same household as the parental participant
* Referred by a health care professional (e.g. physician, midwife, nurse, other professions)

Exclusion Criteria:

* Participation in another study/trial targeting similar outcomes
* Participation in an active smoking cessation programme

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in urinary levels of cotinine in children | At 22 weeks after baseline (Post intervention)
  Change in exposure to second-hand smoke exposure assessed by urinary levels of cotinine
Change from baseline in urinary levels of cotinine in children | At 48 weeks after baseline (Follow-Up)
  Change in exposure to second-hand smoke exposure assessed by urinary levels of cotinine

SECONDARY OUTCOMES:
Change from baseline in protective measures taken by parents to protect children from second-hand smoke exposure | During intervention (week 2-22), post intervention (week 22-23) and follow-up (week 48-49)
  Parents are asked (using a questionnaire) about the measures taken to protect children from second-hand smoke exposure at baseline, during the intervention, postintervention and follow-up. Protective measures assessed include washing hands, smoking outside (including not smoking in the car), changing clothes after smoking). The questionnaire consists of five items (protective measures) with a score ranging from 1 to 5. Score 5 means a better result.

OTHER OUTCOMES:
Acceptance and usability of the app (parent reported outcome) | At 22 weeks after baseline (Post intervention)
  The usability of the app is assessed using the eHealth App Usability Questionnaire (MAUQ). The questionnaire measures usability on three subscales (ease of use, Interface and satisfaction, usefulness). The MAUQ questionnaire consists of 18 items with a score ranging from 1 to 7. Score 7 means a better result.
Acceptance of the app | During the intervention (week 2-22)
  The acceptance of the app is measured by means of dropout rate.
Usability of the app | During the intervention (week 2-22)
  The usability of the app is measured by means of how often and how long the parents use the app.
Number of episodes of airway disease in children | Baseline, at 22 weeks (Post intervention) and at 48 weeks (Follow-Up) after baseline
  Parents are asked to report any event of airway disease (including any type of upper or lower respiratory tract infection; e.g. otitis media, rhinitis, pharyngitis, acute or chronic bronchitis, protracted bacterial bronchitis, chronic cough, pneumonia).
Frequency of inhalant medications or antibiotics required for airway disease in children | Baseline, at 22 weeks (Post intervention) and at 48 weeks (Follow-Up) after baseline
  Parents are asked to report any medical treatment received because of airway disease (includes inhalant drugs, antibiotics, antipyretic medication).
Amount of inhalant medications or antibiotics required for airway disease in children | Baseline, at 22 weeks (Post intervention) and at 48 weeks (Follow-Up) after baseline
  Parents are asked to report any medical treatment received because of airway disease (includes inhalant drugs, antibiotics, antipyretic medication).
Number of episodes of severe airway disease in children requiring hospitalization | Baseline, during the intervention (week 2-22), at 22 weeks (Post intervention) and at 48 weeks (Follow-Up) after baseline
  Parents are asked about any hospitalization because of airway disease.
Change from baseline in parental smoking intensity (number of cigarettes smoked per day) | At 22 weeks (Post intervention) and at 48 weeks (Follow-Up) after baseline
  Parents are asked to report their smoking habits (using a questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias V. Kopp, Prof. Dr., Principal Investigator — Department of Paediatrics, Inselspital, Bern University Hospital, University of Bern, Switzerland; Michael Kaess, Prof. Dr., Principal Investigator — Universitäre Psychiatrische Dienste Bern (UPD), University of Bern, Switzerland
Locations (1):
- Department of Paediatrics, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koch A, Wyssen A, Haupt C, Hammelbeck J, van Dorland HA, Fluck CE, Latzin P, Saner C, Jakob J, Kaess M, Kopp MV. Early Life Intervention in Paediatrics Supported by E-Health (ELIPSE)-a coaching app for parents to reduce obesity and second-hand smoke exposure in children: study protocols for two parallel-group randomised controlled trials. Trials. 2025 Nov 18;26(1):520. doi: 10.1186/s13063-025-09251-5. PMID 41254719